CLINICAL TRIAL: NCT02349412
Title: Randomized Study of Early Palliative Care Integrated With Standard Oncology Care Versus Standard Oncology Care Alone in Patients With Incurable Lung or Non-Colorectal Gastrointestinal Malignancies
Brief Title: Early Palliative Care With Standard Care or Standard Care Alone in Improving Quality of Life of Patients With Incurable Lung or Non-colorectal Gastrointestinal Cancer and Their Family Caregivers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A221303; U10CA037447 (NIH); UG1CA189823 (NIH); NCI-2014-01943 (Registry Identifier: NCI Clinical Trial Reporting Program Office)
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Liver Cancer; Anxiety Disorder; Depression; Small Cell Lung Cancer; Extrahepatic Bile Duct Cancer; Malignant Mesothelioma; Pancreatic Cancer; Esophageal Cancer; Gastric Cancer; Non-small Cell Lung Cancer
MeSH Terms: conditions — Liver Neoplasms; Anxiety Disorders; Depression; Small Cell Lung Carcinoma; Bile Duct Neoplasms; Mesothelioma, Malignant; Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Patients receive early palliative care and standard oncology care. Patients and family caregivers will be asked to complete quality-of-life questionnaires at weeks 6, 12, and 24. Survival follow-up will be every 4 months from week 24 until death or up to 3 years.
  Interventions: Other: Early palliative care
- Arm 2 (Experimental): Patients receive standard oncology care. Patient and family caregiver will be asked to complete self-report questionnaires at weeks 6, 12, and 24. Survival follow-up will be every 4 months from week 24 until death or up to 3 years. Palliative care visit only upon request from attending oncologist(s) or patient/family.
  Interventions: Other: Early palliative care

INTERVENTIONS:
Other: Early palliative care

SUMMARY:
The study intervention consists of the early integration of palliative care services into standard oncology care in an outpatient setting for patients with advanced lung and non-colorectal gastrointestinal malignancies who are not being treated with curative intent. The palliative care services provided to patients randomized to the intervention will be provided by board-certified physicians and/or advanced practice nurses and will focus on the following areas: (1) developing and maintaining the therapeutic relationship with the patients and family caregivers; (2) assessing and treating patient symptoms; (3) providing support and reinforcement of coping with advanced cancer in patients and family caregivers; (4) assessing and enhancing prognostic awareness and illness understanding in patients and family caregivers; (5) assisting with treatment decision-making; and (6) end-of-life care planning.

DETAILED DESCRIPTION:
There will be about 400 patients enrolled in this intervention study and there will be about 300 family caregivers enrolled as well. This study will consist of two study groups as previously described. The effects of the early involvement of the palliative care team will be compared to the usual approach of receiving care mostly from the cancer treatment team. The stratification factors include tumor type (lung vs. esophageal/gastric vs. hepatic/biliary/pancreatic) and family care giver participation (yes vs. no). Patients will be on this study for as long as they receive care. Institutions must have an outpatient palliative care clinic that meets the study site requirements as defined in the protocol. The outpatient clinic leadership must include a physician and/or advanced practice nurses board certified in palliative care. The primary and secondary endpoints are described below.

Primary Endpoint:

To determine the efficacy of early integrated palliative care on patient reported quality of life at 12 weeks using the FACT in patients with newly diagnosed incurable lung or non-colorectal gastrointestinal cancer

Secondary Endpoints:

* To determine the efficacy of early integrated palliative care on other patient reported outcomes in patients with newly diagnosed incurable lung or non-colorectal gastrointestinal cancer, by assessing the endpoints defined in the protocol
* To determine the efficacy of early integrated palliative care on family caregiver reported outcomes in those newly diagnosed incurable lung or non-colorectal gastrointestinal cancer, by assessing the endpoints defined in the protocol
* To assess the impact of early integrated palliative care on the quality of end-of-life care and resource utilization in patients with newly diagnosed incurable lung or non-colorectal gastrointestinal cancer by assessing the endpoints defined in the protocol
* To determine concordance between patient and family caregiver report of prognosis/ curability

ELIGIBILITY:
Study Patient Participant Eligibility Requirements:

1. Documentation of Disease: Confirmed advanced lung cancer (NSCLC, small cell lung cancer, or mesothelioma) or non-colorectal GI cancer (esophageal, gastric, hepatic, biliary, or pancreatic) not being treated with curative intent.
2. Informed of diagnosis of incurable disease within the previous 8 weeks.
3. Age ≥ 18 years
4. ECOG Performance Status 0-2
5. Ability to read and respond to questions in English or able to complete questions with minimal assistance required from an interpreter or family member.
6. Planning to receive all medical care for cancer at the enrolling institution.
7. Participants must be under the care of an oncologist, but their current plan may or may not include chemotherapy or other forms of tumor-directed therapies.

Study Family Caregiver Participant Eligibility Requirements:

1. Relative or friend who is identified by the patient participant who plans to regularly accompany the patient to the majority of their clinic visits.
2. Family caregiver must live with the patient or have in-person contact with him or her at least twice per week.
3. Ability to read and respond to questions in English or able to complete questions with minimal assistance required from an interpreter or family member.
4. Age ≥ 18 years

Note: An eligible patient may participate in this trial without an eligible family caregiver being registered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Temel, MD, Study Chair — Massachusetts General Hospital
Locations (23):
- United States (23):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Temel JS, Sloan J, Zemla T, Greer JA, Jackson VA, El-Jawahri A, Kamdar M, Kamal A, Blinderman CD, Strand J, Zylla D, Daugherty C, Furqan M, Obel J, Razaq M, Roeland EJ, Loprinzi C. Multisite, Randomized Trial of Early Integrated Palliative and Oncology Care in Patients with Advanced Lung and Gastrointestinal Cancer: Alliance A221303. J Palliat Med. 2020 Jul;23(7):922-929. doi: 10.1089/jpm.2019.0377. Epub 2020 Feb 7. PMID 32031887
- [Derived] Jacobs JM, Shaffer KM, Nipp RD, Fishbein JN, MacDonald J, El-Jawahri A, Pirl WF, Jackson VA, Park ER, Temel JS, Greer JA. Distress is Interdependent in Patients and Caregivers with Newly Diagnosed Incurable Cancers. Ann Behav Med. 2017 Aug;51(4):519-531. doi: 10.1007/s12160-017-9875-3. PMID 28097515
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (Early Palliative Care): Patients receive early palliative care and standard oncology care. Patients and family caregivers will be asked to complete quality-of-life questionnaires at weeks 6, 12, and 24. Survival follow-up will be every 4 months from week 24 until death or up to 3 years.
- Arm 2 (Usual Care): Patients receive standard oncology care. Patient and family caregiver will be asked to complete self-report questionnaires at weeks 6, 12, and 24. Survival follow-up will be every 4 months from week 24 until death or up to 3 years. Palliative care visit only upon request from attending oncologist(s) or patient/family.
Period: Overall Study
Arm/Group | Arm 1 (Early Palliative Care) | Arm 2 (Usual Care)
Started | 202 | 203
Completed Week-12 QOL Assessment Measure | 92 | 101
Completed Week-24 QOL Assessment Measure | 68 | 80
Completed | 195 | 196
Not Completed | 7 | 7
Not completed — Withdrawal by Subject | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Early Palliative Care) | Arm 2 (Usual Care) | Total
Number analyzed (Participants) | 195 | 196 | 391
Age, Continuous [Mean (Full Range); unit: years] | 65.5 [35 to 97] | 65.0 [34 to 92] | 65.2 [34 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 89 | 170
  Male | 114 | 107 | 221
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 9 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 24 | 22 | 46
  White | 148 | 155 | 303
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 9 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 195 | 196 | 391
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 47 | 41 | 88
    1 | 108 | 127 | 235
    2 | 40 | 28 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life (QOL) From Baseline to Week 12 Per the Functional Assessment of Cancer Therapy-General (FACT-G)
Description: Quality of Life (QOL) was measured using the Functional Assessment of Cancer Therapy-General (FACT-G) on a 0-108 scale, with lower scores corresponding to worse overall QOL and higher scores corresponding to better overall QOL. Change from baseline to week-12 was calculated by subtracting the baseline scores from the scores at week-12. Higher scores on FACT-G indicate better QOL.
Time Frame: Up to 12 weeks
Population: Only participants with available data on the individual study measure at baseline and 12 weeks were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 (Early Palliative Care) | Arm 2 (Usual Care)
Number analyzed (Participants) | 92 | 101
units on a scale | 3.35 (14.7) | 0.12 (12.7)
Statistical Analysis 1: Comparison: Arm 1 (Early Palliative Care) vs Arm 2 (Usual Care); Test type: Superiority; p = 0.104, ANCOVA; Statistical Method: Available Case ANCOVA Model adjusting for baseline FACT-G score; Mean Difference (Final Values) = 3.23, 95% CI 2-sided [-0.67 to 7.13]

2. Secondary Outcome: Change in Quality of Life (QOL) From Baseline to Week 24 Per the Functional Assessment of Cancer Therapy-General (FACT-G)
Description: Quality of Life (QOL) was measured using the Functional Assessment of Cancer Therapy-General (FACT-G) on a 0-108 scale, with lower scores corresponding to worse overall QOL and higher scores corresponding to better overall QOL. Change from baseline to week-24 was calculated by subtracting the baseline scores from the scores at week-24. Higher scores on FACT-G indicate better QOL.
Time Frame: Up to 24 weeks
Population: Only participants with available data on the individual study measure at baseline and 24 weeks were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 (Early Palliative Care) | Arm 2 (Usual Care)
Number analyzed (Participants) | 68 | 80
units on a scale | 3.80 (15.3) | 0.69 (13.3)
Statistical Analysis 1: Comparison: Arm 1 (Early Palliative Care) vs Arm 2 (Usual Care); Test type: Superiority; p = 0.188, ANCOVA; Statistical Method: Available Case ANCOVA Model adjusting for baseline FACT-G score; Mean Difference (Final Values) = 3.12, 95% CI 2-sided [-1.54 to 7.77]

3. Secondary Outcome: Change in Quality of Life (QOL) From Baseline to Week 12 Per the Hospital Anxiety and Depression Scale (HADS) - Depression
Description: Quality of Life (QOL) was measured using the Hospital Anxiety and Depression Scale (HADS) - Depression on a 0-21 scale, with lower scores corresponding to lower depression and higher scores corresponding to higher depression. Change from baseline to week-12 was calculated by subtracting the baseline scores from the scores at week-12. Lower scores on the HADS-Depression indicate less depression symptoms.
Time Frame: Up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 (Early Palliative Care) | Arm 2 (Usual Care)
Number analyzed (Participants) | 100 | 112
units on a scale | 0.54 (4.0) | 0.46 (3.6)
Statistical Analysis 1: Comparison: Arm 1 (Early Palliative Care) vs Arm 2 (Usual Care); Test type: Superiority; p = 0.884, ANCOVA; Statistical Method: Available Case ANCOVA Model adjusting for baseline HADS-Depression score; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.94 to 2.09]

4. Secondary Outcome: Change in Quality of Life (QOL) From Baseline to Week 12 Per the Hospital Anxiety and Depression Scale (HADS) - Anxiety
Description: Quality of Life (QOL) was measured using the Hospital Anxiety and Depression Scale (HADS) - Anxiety on a 0-21 scale, with lower scores corresponding to lower anxiety and higher scores corresponding to higher anxiety. Change from baseline to week-12 was calculated by subtracting the baseline scores from the scores at week-12. Lower scores on the HADS-Anxiety indicate less anxiety symptoms.
Time Frame: Up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 (Early Palliative Care) | Arm 2 (Usual Care)
Number analyzed (Participants) | 100 | 111
units on a scale | -1.13 (2.7) | -0.32 (2.8)
Statistical Analysis 1: Comparison: Arm 1 (Early Palliative Care) vs Arm 2 (Usual Care); Test type: Superiority; p = 0.033, ANCOVA; Statistical Method: Available Case ANCOVA Model adjusting for baseline HADS-Anxiety score; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.54 to -0.07]

5. Secondary Outcome: Prognostic Understanding at Week-12 as Measured by "Have You and Your Oncologist Discussed Any Particular Wishes About the Care You Would Want to Receive if You Were Dying?" Question on the Prognosis and Treatment Perceptions Questionnaire
Description: Prognostic Understanding at Week-12 as measured by Prognosis and Treatment Perceptions Questionnaire: "Have you and your oncologist discussed any particular wishes about the care you would want to receive if you were dying?" responses at Week-12 are reported below.
Time Frame: Up to 12 weeks
Population: Only participants with available data on the individual study measure at week 12 were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Early Palliative Care) | Arm 2 (Usual Care)
Number analyzed (Participants) | 99 | 110
Participants
  Yes | 30 | 16
  No | 69 | 94
Statistical Analysis 1: Comparison: Arm 1 (Early Palliative Care) vs Arm 2 (Usual Care); Test type: Superiority; p = 0.006, Chi-squared

6. Secondary Outcome: Change in QOL on the SF-36 Over Time
Time Frame: Up to 3 years
Reporting Status: Not Posted

7. Secondary Outcome: Rate of Referral, Enrollment and Length of Stay on Hospice
Time Frame: Up to 3 years
Reporting Status: Not Posted

8. Secondary Outcome: Location of Death
Time Frame: Up to 3 years
Reporting Status: Not Posted

9. Secondary Outcome: Number of Hospital and Intensive Care Unit (ICU) Admissions and Days
Time Frame: Up to 3 years
Reporting Status: Not Posted

10. Secondary Outcome: Chemotherapy and Radiation Administration
Time Frame: Up to 3 years
Reporting Status: Not Posted

11. Secondary Outcome: Overall Survival
Time Frame: Up to 3 years
Reporting Status: Not Posted

12. Secondary Outcome: Concordance Between Patient and Family Caregiver Report of Prognosis/Curability
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study.
Description: Adverse events were not collected for this study.
Arm/Group | Arm 1 (Early Palliative Care) | Arm 2 (Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT02349412/Prot_SAP_ICF_000.pdf